CLINICAL TRIAL: NCT04154137
Title: Prevalence of Self-reported Non-celiac Wheat Sensitivity (NCWS) in Patients Undergoing Digestive Endoscopy
Brief Title: Self-reported Non-celiac Wheat Sensitivity (NCWS) in Patients Undergoing Digestive Endoscopy
Status: Completed | Type: Observational
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Pasquale Mansueto, Clinical Professor, University of Palermo
Other Study IDs: ACPM23
Record Dates: First submitted 2019-11-04; First posted 2019-11-06 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Non-celiac Wheat Sensitivity
Keywords: non-celiac wheat sensitivity; celiac disease; wheat allergy
MeSH Terms: conditions — Celiac Disease; Wheat Hypersensitivity | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing digestive endoscopy: All the patients, age ranged from 18 to 90 years, referred to Digestive Endoscopy Outpatients Clinic of the Department of Gastroenterology of the University Hospital "Paolo Giaccone" of Palermo, Italy
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Enrolled patients will fill out a modified version of a previously validated written questionnaire, including two different sections. The first comprises basic demographic information, including age, sex and ethnicity, and a screening section for symptoms consistent with irritable bowel syndrome (IBS) in accordance with the Rome III criteria, also including their past gastrointestinal, allergic and psychiatric history. The second section enquires for self-reported gluten-related symptoms. Participants will be also asked for their use of a gluten-free diet and if they had seen a healthcare professional for their symptoms. A reported diagnosis of celiac disease and wheat allergy in the population group is defined by those who had a doctor diagnosis of celiac disease and wheat allergy and are also taking a gluten-free diet.

SUMMARY:
Self-reported food hypersensitivity is common, particularly in women, with a reported prevalence of about 20% in the UK community. A wide range of gastrointestinal and systemic symptoms may be experienced related to consumption of the intolerant food(s). In addition, patients demonstrate considerably more generalized subjective health complaints in comparison with healthy controls. In this context, it has been reported that a consistent percentage of the general population consider themselves to be suffering from problems caused by wheat and/or gluten ingestion, even though they do not have celiac disease or wheat allergy. This clinical condition has been named non-celiac gluten sensitivity' (NCGS). In a previous paper the investigators suggested the term 'non-celiac wheat sensitivity' (NCWS), since it is not known what component of wheat causes the symptoms in NCGS patients, and the investigators also showed that these patients had a high frequency of coexistent multiple food hypersensitivity. In a previous study, the investigators demonstrated, in a population of teenagers, a frequency of self-reported NCWS of about 12%; the frequency of GFD use was 2.9%, which was much higher than the percentage of known CD in the same population (1.26%). The aims of this study were 1) to determine the prevalence of self-perceived wheat and/or gluten-sensitivity in patients undergoing digestive endoscopy, irrespective to the motivations of the test, and 2) to evaluate the demographic and clinical differences between patients self-reporting wheat and/or gluten sensitivity and patients not reporting food hypersensitivity.

DETAILED DESCRIPTION:
Self-reported food hypersensitivity is common, particularly in women, with a reported prevalence of about 20% in the UK community. A wide range of gastrointestinal and systemic symptoms may be experienced related to consumption of the intolerant food(s). In addition, patients demonstrate considerably more generalized subjective health complaints in comparison with healthy controls. In this context, it has been reported that a consistent percentage of the general population consider themselves to be suffering from problems caused by wheat and/or gluten ingestion, even though they do not have celiac disease or wheat allergy. This clinical condition has been named non-celiac gluten sensitivity' (NCGS). In a previous paper the investigators suggested the term 'non-celiac wheat sensitivity' (NCWS), since it is not known what component of wheat causes the symptoms in NCGS patients, and the investigators also showed that these patients had a high frequency of coexistent multiple food hypersensitivity. The clinical picture of NCWS is characterized by combined gastrointestinal (bloating, abdominal pain, diarrhea and/or constipation, nausea, epigastric pain, gastroesophageal reflux, aphthous stomatitis) and extra-intestinal and/or systemic manifestations (headache, depression, anxiety, 'foggy mind,' tiredness, dermatitis or skin rash, fibromyalgia-like joint/muscle pain, leg or arm numbness, and anemia). To our knowledge, there are few studies which assessed the prevalence of self-reported wheat and/or gluten-related symptoms in the community and analyze diagnostic outcomes in those referred to secondary gastrointestinal care. In one of these, performed in UK, the authors shown that gluten-related symptoms are self-reported by 13% of the population, with 3.7% consuming a gluten-free diet, despite only 0.8% being aware that they have a formal diagnosis of celiac disease. In this study individuals self-reporting gluten-related symptoms were predominantly female, reported an association with IBS, and experienced both intestinal and extraintestinal symptoms on gluten ingestion. Of those patients presenting to the gastroenterology department, the majority do not have CD but NCWS. In another study, the investigators demonstrated, in a population of teenagers, a frequency of self-reported NCWS of about 12%; the frequency of GFD use was 2.9%, which was much higher than the percentage of known CD in the same population (1.26%). The aims of this study were 1) to determine the prevalence of self-perceived wheat and/or gluten-sensitivity in patients undergoing digestive endoscopy, irrespective to the motivations of the test, and 2) to evaluate the demographic and clinical differences between patients self-reporting wheat and/or gluten sensitivity and patients not reporting food hypersensitivity.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing digestive endoscopic investigations, irrespective to the motivations of the test.

Exclusion Criteria:

* None

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study will include patients undergoing digestive endoscopy (i.e. esophagogastroduodenoscopy, pancolonscopy and proctoscopy), at the Digestive Endoscopy Outpatients Clinic of the Department of Gastroenterology of the University Hospital "Paolo Giaccone" of Palermo, Italy, between January 2017 and January 2020.
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Self-perceived wheat and/or gluten-sensitivity in patients undergoing digestive endoscopy. | January 2017 to January 2020
  Prevalence of self-perceived wheat and/or gluten-sensitivity in patients undergoing digestive endoscopy by using an ad hoc questionnaire.

SECONDARY OUTCOMES:
Differences between patients self-reporting wheat and/or gluten sensitivity and patients not reporting food hypersensitivity. | January 2017 to January 2020
  Demographic and clinical differences between patients self-reporting wheat and/or gluten sensitivity and patients not reporting food hypersensitivity.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Carroccio, PHD, Study Director — University of Palermo
Locations (3):
- Italy (3):
  - Digestive Endoscopy Outpatients Clinic of the Department of Gastroenterology of the University Hospital "Paolo Giaccone", Palermo, PA
  - Internal Medicine Division of the "Cervello-Villa Sofia" Hospital, Palermo, PA
  - Department of Internal Medicine, University Hospital of Palermo, Palermo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Carroccio A, Mansueto P, Iacono G, Soresi M, D'Alcamo A, Cavataio F, Brusca I, Florena AM, Ambrosiano G, Seidita A, Pirrone G, Rini GB. Non-celiac wheat sensitivity diagnosed by double-blind placebo-controlled challenge: exploring a new clinical entity. Am J Gastroenterol. 2012 Dec;107(12):1898-906; quiz 1907. doi: 10.1038/ajg.2012.236. Epub 2012 Jul 24. PMID 22825366
- [Result] Mansueto P, Seidita A, D'Alcamo A, Carroccio A. Non-celiac gluten sensitivity: literature review. J Am Coll Nutr. 2014;33(1):39-54. doi: 10.1080/07315724.2014.869996. PMID 24533607
- [Result] Carroccio A, Rini G, Mansueto P. Non-celiac wheat sensitivity is a more appropriate label than non-celiac gluten sensitivity. Gastroenterology. 2014 Jan;146(1):320-1. doi: 10.1053/j.gastro.2013.08.061. Epub 2013 Nov 22. No abstract available. PMID 24275240
- [Result] Carroccio A, D'Alcamo A, Mansueto P. Nonceliac wheat sensitivity in the context of multiple food hypersensitivity: new data from confocal endomicroscopy. Gastroenterology. 2015 Mar;148(3):666-7. doi: 10.1053/j.gastro.2014.11.047. Epub 2015 Jan 24. No abstract available. PMID 25625764
- [Result] Carroccio A, Soresi M, D'Alcamo A, Sciume C, Iacono G, Geraci G, Brusca I, Seidita A, Adragna F, Carta M, Mansueto P. Risk of low bone mineral density and low body mass index in patients with non-celiac wheat-sensitivity: a prospective observation study. BMC Med. 2014 Nov 28;12:230. doi: 10.1186/s12916-014-0230-2. PMID 25430806
- [Result] Mansueto P, Seidita A, D'Alcamo A, Carroccio A. Role of FODMAPs in Patients With Irritable Bowel Syndrome. Nutr Clin Pract. 2015 Oct;30(5):665-82. doi: 10.1177/0884533615569886. Epub 2015 Feb 18. PMID 25694210
- [Result] Young E, Stoneham MD, Petruckevitch A, Barton J, Rona R. A population study of food intolerance. Lancet. 1994 May 7;343(8906):1127-30. doi: 10.1016/s0140-6736(94)90234-8. PMID 7910231
- [Result] Aziz I, Lewis NR, Hadjivassiliou M, Winfield SN, Rugg N, Kelsall A, Newrick L, Sanders DS. A UK study assessing the population prevalence of self-reported gluten sensitivity and referral characteristics to secondary care. Eur J Gastroenterol Hepatol. 2014 Jan;26(1):33-9. doi: 10.1097/01.meg.0000435546.87251.f7. PMID 24216570
- [Result] Sanders DS, Patel D, Stephenson TJ, Ward AM, McCloskey EV, Hadjivassiliou M, Lobo AJ. A primary care cross-sectional study of undiagnosed adult coeliac disease. Eur J Gastroenterol Hepatol. 2003 Apr;15(4):407-13. doi: 10.1097/00042737-200304000-00012. PMID 12655262
- [Derived] Mansueto P, Soresi M, Peralta S, Perricone S, La Blasca F, Sichera R, Giambalvo O, Carroccio A. Self-reported nonceliac wheat sensitivity in an outpatient digestive endoscopy center: high frequency but insufficient medical approach. Eur J Gastroenterol Hepatol. 2021 Dec 1;33(1S Suppl 1):e789-e795. doi: 10.1097/MEG.0000000000002257. PMID 34334709